CLINICAL TRIAL: NCT06478004
Title: Direct Resin Composite Restoration of Primary Anterior Teeth Using Custom 3D Printed Templates: A 12-Month Parallel Randomized Controlled Clinical Trial
Brief Title: Direct Resin Composite Restoration of Primary Anterior Teeth Using Custom 3D Printed Templates
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Kamal Yassa, Lecturer in Paediatric and Community Dentistry Department, Faculty of Dentistry, Minia University, Minia, Egypt., Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #841/2023
Record Dates: First submitted 2024-06-15; First posted 2024-06-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Primary Teeth
Keywords: Early childhood caries; Strip Crown; 3D Printing

STUDY DESIGN:
Intervention Model Description: Single-center, prospective randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct resin composite with the help of custom 3D printed templates (Experimental): Directly restoring carious primary anterior teeth with resin composite with the help of custom 3D printed templates obtained from digitally waxed-up patients' dental models.
  Interventions: Other: Direct composite restoration of carious primary anterior teeth using custom 3D printed templates
- Direct resin composite using conventional strip crowns. (Active Comparator): Directly restoring carious primary anterior teeth with resin composite using conventional strip crowns.
  Interventions: Other: Direct composite restoration of carious primary anterior teeth using conventional strip crowns

INTERVENTIONS:
Other: Direct composite restoration of carious primary anterior teeth using custom 3D printed templates — A patient dental model is acquired by digital scan then digital waxing-up is performed using the Exocad software to 3D print clear templates for direct composite resin restoration.
  Arms: Direct resin composite with the help of custom 3D printed templates
Other: Direct composite restoration of carious primary anterior teeth using conventional strip crowns — Direct composite resin restoration using celluloid crown forms
  Arms: Direct resin composite using conventional strip crowns.

SUMMARY:
Esthetic restoration of primary anterior teeth is challenging. Aim of the study: Evaluation of the 12-month clinical performance of direct resin composite restoration of carious vital primary anterior teeth using custom 3D printed templates compared to conventional strip crowns. Subjects and methods: A parallel arms randomized controlled clinical trial was performed in which 98 carious vital primary anterior teeth in 32 children were directly restored with resin composite either with the help of custom 3D printed templates (Group: A) or strip crowns (Group: B). Restorations were assessed for surface luster, anatomical form, material fracture, marginal adaptation, and periodontal response using the revised FDI criteria on three occasions; a week after placement (T0), after six months (T1), and after twelve months (T2). Comparisons between groups were evaluated. A statistically significant level was considered when p value less than or equal 0.05. The tooth was the unit of analysis.

DETAILED DESCRIPTION:
The present study is a single-center randomized controlled clinical trial with 1:1 allocation ratio. This trial entailed directly restoring carious primary anterior teeth with resin composite either with the help of custom 3D printed templates obtained from digitally waxed-up patients' dental models (Group: A) or conventional strip crowns (Group: B). Restorations were assessed for clinical performance on three occasions; postoperatively (T0), after six months (T1), and after twelve months (T2).

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least two vital carious primary maxillary incisors.
* Teeth had at least two carious surfaces requiring complete coronal restoration.

Exclusion Criteria:

* Children with malocclusion or parafunctional oral habits
* Teeth beyond restoration.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Surface luster | On three occasions; a week after placement (T0), at six months (T1), and at twelve months (T2)
  Assessment according to the revised clinical criteria for the evaluation of direct and indirect restorations of the World Dental Federation (FDI), Each criterion was scored according to a five-step grading of the restoration that was then dichotomized into "acceptable" (for scores 1, 2&3) and "not acceptable" (for scores 4&5)
Anatomical form | On three occasions; a week after placement (T0), at six months (T1), and at twelve months (T2)
  Assessment according to the revised clinical criteria for the evaluation of direct and indirect restorations of the World Dental Federation (FDI), Each criterion was scored according to a five-step grading of the restoration that was then dichotomized into "acceptable" (for scores 1, 2&3) and "not acceptable" (for scores 4&5)
Material fracture | On three occasions; a week after placement (T0), at six months (T1), and at twelve months (T2)
  Assessment according to the revised clinical criteria for the evaluation of direct and indirect restorations of the World Dental Federation (FDI), Each criterion was scored according to a five-step grading of the restoration that was then dichotomized into "acceptable" (for scores 1, 2&3) and "not acceptable" (for scores 4&5)
Marginal adaptation | On three occasions; a week after placement (T0), at six months (T1), and at twelve months (T2)
  Assessment according to the revised clinical criteria for the evaluation of direct and indirect restorations of the World Dental Federation (FDI), Each criterion was scored according to a five-step grading of the restoration that was then dichotomized into "acceptable" (for scores 1, 2&3) and "not acceptable" (for scores 4&5)
Periodontal response | On three occasions; a week after placement (T0), at six months (T1), and at twelve months (T2)
  Assessment according to the revised clinical criteria for the evaluation of direct and indirect restorations of the World Dental Federation (FDI), Each criterion was scored according to a five-step grading of the restoration that was then dichotomized into "acceptable" (for scores 1, 2&3) and "not acceptable" (for scores 4&5)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Yassa, Doctor, Principal Investigator — Faculty of Dentistry, Minia University, Minia, Egypt.
Locations (1):
- Faculty of Dentistry, Minia University, Minya, Egypt